CLINICAL TRIAL: NCT05606614
Title: An Open-label Phase 1/2/3 Study Consisting of a Phase 1/2 Safety and Dose-escalation and Phase 3 Dose-expansion Study to Evaluate Safety and Efficacy of a Single Intrathecal Administration of TSHA-102, an AAV9-Delivered Gene Therapy in Females With Rett Syndrome
Brief Title: A Phase 1/2/3 Study of TSHA-102 Gene Therapy in Females With Rett Syndrome (REVEAL Pivotal Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taysha Gene Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TSHA-102-CL-101
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Neurodevelopmental disorder; Rett; MECP2; AAV9; Typical Rett Syndrome; Classic Rett Syndrome; RTT; Rett Disorder; Retts; MECP2-Related Disorder; Gene Therapy; Intrathecal Administration; Genetic Diseases, X-Linked; Nervous System Diseases; Developmental Regression; TSHA-102; miRARE; Self-complementary Vector; Neurologic Manifestations; Intellectual Disability; Pathologic Process; X-Linked Intellectual Disability; Congenital, Hereditary, and Neonatal Diseases and Abnormalities
MeSH Terms: conditions — Rett Syndrome; Neurodevelopmental Disorders; Genetic Diseases, X-Linked; Nervous System Diseases; Neurologic Manifestations; Intellectual Disability; Pathologic Processes; X-Linked Intellectual Disability; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Intervention Model Description: The study treatment will be delivered via intrathecal (IT) injection.
Who Masked: Outcomes Assessor
Masking Description: Central raters assessing the gain or regain of a developmental milestone from videos are blinded to the timing of each video.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A Cohort 1 (Experimental): TSHA-102 Dose Level 1: 5.7×10¹⁴ total vector genomes (vg). Participants receive a single intrathecal (IT) administration of TSHA-102 at Dose Level 1 (fully enrolled, 2 participants).
  Interventions: Genetic: TSHA-102
- Part A Cohort 2 (Experimental): TSHA-102 Dose Level 2: 1.0×10¹⁵ total vector genomes (vg)
  Participants receive a single intrathecal (IT) administration of TSHA-102 at Dose Level 2 (fully enrolled, 4 participants).
  Interventions: Genetic: TSHA-102
- Part B Pivotal Cohort (Experimental): TSHA-102 at Selected Dose (Dose Level 2): 1.0 × 10¹⁵ total vector genomes (vg)
  Participants receive a single intrathecal (IT) administration of TSHA-102 at Dose Level 2 (1.0 × 10¹⁵).
  Interventions: Genetic: TSHA-102

INTERVENTIONS:
Genetic: TSHA-102 — TSHA-102 is a recombinant, non-replicating, self-complementary AAV9 (scAAV9) vector encoding for the miniMECP2 gene. TSHA-102 is a one-time intrathecal (IT) administration.

SUMMARY:
The primary objectives of this study are to evaluate the safety of a single intrathecal (IT) dose of TSHA-102 in females with typical Rett syndrome, to select the TSHA-102 dose with the best benefit/risk profile based on the totality of safety and efficacy data and to evaluate the efficacy and safety of TSHA-102 at the selected dose.

DETAILED DESCRIPTION:
REVEAL Part A (Phase 1/2) is an open-label safety and dose-finding study designed to evaluate the safety and preliminary efficacy of two dose levels of TSHA-102 to establish initial safety of TSHA-102 and select a safe and efficacious dose for further evaluation. Enrollment of 6 participants in Part A is complete.

REVEAL Part B (Phase 3) will evaluate the efficacy and safety of TSHA-102 at the dose level 2 determined in Part A in 15 females ages 6 to <22 years with typical Rett syndrome. TSHA-102 is designed to target the genetic root cause of Rett syndrome by regulating the expression of MECP2 in cells.

Each participant will be followed for the observation period of 5 years after TSHA-102 administration in Part A and B.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 12 and <22 in Part A (closed) and females between the ages of 6 and <22 in Part B (pivotal cohort).
* Participant has a clinical diagnosis of classic/typical Rett syndrome with a documented pathogenic mutation of the methyl-CpG-binding protein 2 (MECP2) gene that results in loss of gene function.
* Participants must be willing to receive blood or blood products for the treatment of an AE if medically needed.
* Participants and parent/caregiver must agree to reside within easy access to the study site prior to the baseline visit and at least 3 months after TSHA-102 treatment

Exclusion Criteria:

* Participant has another neurodevelopmental disorder independent of the MECP2 loss-of-function mutation, or any other genetic syndrome with a progressive course.
* Participant has a history of brain injury that causes neurological problems or had grossly abnormal psychomotor development in the first 6 months of life.
* Participant has a diagnosis of atypical Rett syndrome or a MECP2 gene mutation that does not cause Rett syndrome.
* Participant requires invasive ventilatory support.

Note: Other protocol defined inclusion/exclusion criteria may apply

Ages: 6 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability of TSHA-102 | Baseline through Week 52
  Proportions of participants experiencing any treatment-emergent adverse events (AEs) and serious adverse events (SAEs)
Part B: Efficacy of TSHA-102 | Baseline through Week 52
  Change from baseline in percentage of participants who gain or regain any one or more of the 28 items from the Developmental Milestones Assessment (DMA), which are video recorded and scored by independent, blinded central raters.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, M.D., Study Director — Taysha Gene Therapies
Locations (6):
- United States (5):
  - UC San Diego, La Jolla, California
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St. Louis, St Louis, Missouri
  - UT Southwestern Children's Medical Center, Dallas, Texas
- CHU St. Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jagadeeswaran I, Oh J, Sinnett SE. Preclinical Milestones in MECP2 Gene Transfer for Treating Rett Syndrome. Dev Neurosci. 2025;47(2):147-156. doi: 10.1159/000539267. Epub 2024 May 9. PMID 38723617
- [Derived] Sadhu C, Lyons C, Oh J, Jagadeeswaran I, Gray SJ, Sinnett SE. The Efficacy of a Human-Ready miniMECP2 Gene Therapy in a Pre-Clinical Model of Rett Syndrome. Genes (Basel). 2023 Dec 24;15(1):31. doi: 10.3390/genes15010031. PMID 38254921